CLINICAL TRIAL: NCT05038683
Title: Holbæk Obesity Treatment (HOT) Versus Conventional Obesity Treatment (COT) in Children With Overweight or Obesity. An Investigator-initiated, Multi-center, Randomized, Parallel Group, Clinical Superiority Trial With Blinded Outcome Assessment. HOT Versus COT Trial.
Brief Title: Holbæk Obesity Treatment (HOT) Versus Conventional Obesity Treatment (COT) in Children With Overweight or Obesity.
Acronym: HOT vs COT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Holbaek Sygehus (Other)
Collaborators: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); University of Copenhagen (Other); Statens Serum Institut (Other); University of Florida (Other); Leeds Beckett University (Other); University of Minnesota (Other); Hebrew University of Jerusalem (Other); Frederiksberg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HOT vs COT trial
Record Dates: First submitted 2021-09-07; First posted 2021-09-09 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Childhood Overweight and Obesity
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the interventions, it will not be possible to blind the healthcare providers administering the interventions. We will attempt to blind the participants by not informing them about which intervention group we consider experimental and which group we consider control. However, the participants included in HOT will be governed by a digital solution where Dr. Holm will be identifiable and thus revealing the HOT. In all other aspects of the trial, we will employ blinding, incl. outcome assessment. Statisticians, and investigators drawing conclusions will be fully blinded. We will conduct the statistical analyses with the intervention groups coded as eg. 'A' and 'B'. The steering committee will write two abstracts while the blinding is intact; one assuming the experimental intervention group is 'A' and the control intervention group is 'B', and one assuming the opposite. After these two abstracts have both obtained consensus, the code will be broken.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HOT (Experimental): Holbæk Obesity Treatment
  Interventions: Behavioral: Holbæk Obesity Treatment
- COT (Active Comparator): Conventional Obesity Treatment
  Interventions: Behavioral: Conventional Obesity Treatment

INTERVENTIONS:
Behavioral: Holbæk Obesity Treatment — Obesity is a chronic, progressive, severe, recidivistic, and complex disease, which mandates that children and adolescents with overweight or obesity have access to a professional medical healthcare service as other pediatric chronic diseases, implying a lifelong course of treatment. The HOT method is further based on the physiological insight into the endocrine regulation of fat mass; especially on how the body adapts when it is challenged by weight loss. These insights include an understanding where the body shifts into an energy-preserving mode when the individual is initiating weight-reducing actions, such as a reduced caloric intake or an increased level of physical activity, which has numerous impacts on communication and pedagogy.
  HOT is administered by healthcare nurses and dietitians at healthcare centers in Danish municipalities. Each treatment will be conducted as face-to-face sessions totalling a range of six to 12 hours for 12 months.
  Arms: HOT
Behavioral: Conventional Obesity Treatment — Obesity is viewed as a chronic disease that is ultimately thought to result from an imbalance between energy intake and energy expenditure. However, multiple factors, both environmental and genetic, are thought to influence the disease as well. As obesity reflects energy imbalances, the treatment plan should be designed to induce a slightly negative energy balance by focusing on diet, physical activity, and inactivity through behavior change. Taking one step at a time, will in the end lead to the same energy balance result (i.e. weight loss) and will be more sustainable for the participant whose motivation is absolutely pivotal in this process.
  COT is administered by healthcare nurses and dietitians at healthcare centers in Danish municipalities. Each treatment will be conducted as face-to-face sessions totalling a range of six to 12 hours for 12 months.
  Arms: COT

SUMMARY:
The HOT versus COT trial aims to compare the effectiveness of two different lifestyle interventions for treatment of childhood overweight and obesity with the purpose of informing future clinical practice guidelines within this field. The aim is to conduct this investigation in an optimal trial design with the lowest possible risk of bias.

DETAILED DESCRIPTION:
Obesity is a chronic, progressive, and severe disease that compromises growth, development, and the general health and well-being of children, adolescents, and adults all around the globe. Current treatment within this field varies considerably, but the prevailing concept is that treatment should be lifelong with a focus on implementing and maintaining changes regarding diet, physical activity, sedentary behavior, sleep, etc. The Holbæk Obesity Treatment (HOT) is built on the understanding that obesity is a complex chronic disease regulated by a neuroendocrine system, where weight-reducing actions initiate counteractive mechanisms to defend fat mass. Conventional obesity treatment (COT) is based on a view that obesity results from energy imbalances and focuses on motivation, few changes at a time, and a narrative approach towards healthy energy intake and physical activity. These two approaches represent fundamentally different treatments of overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obesity defined as BMI corresponding to or above the 90th percentile for age and sex (International Obesity Task Force cut-offs).
* Age six to < 12 years at enrolment.
* Signed informed consent from both parents or legal guardians.

Exclusion Criteria:

* Participation in multidisciplinary obesity treatment (i.e. treatment involving more than one type of healthcare profession) within the past 12 months.
* Having a sibling already enrolled in the HOT versus COT trial.
* Both parents or legal guardians unable to communicate in Danish (written or oral).
* Child unable to communicate in Danish (oral).
* Current or previous clinical diagnosis of either anorexia or bulimia according to ICD-10.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 554 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
BMI SDS | End of intervention (12 months)
  BMI SDS assessed according to the International Obesity Task Force cut-offs.
Quality of life (PedsQL) | End of intervention (12 months)
  Quality of life assessed by Pediatric Quality of Life Inventory (PedsQL)

OTHER OUTCOMES:
Symptoms of depression and anxiety | End of intervention (12 months)
  Symptoms of depression and anxiety assessed with the questionnaire RCADS.
Serious adverse events (SAE) | End of intervention (12 months)
  Proportion of participants with one or more SAEs defined as any adverse event that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, or results in persistent or significant disability or incapacity.
Anorexia or bulimia | End of intervention (12 months)
  Proportion of participants with a clinical diagnosis of anorexia or bulimia
School absence | End of intervention (12 months)
  Number of days absent from kindergarten and school (excluding holidays).
Body composition | End of intervention (12 months)
  Body composition, defined as % body fat by using bioelectrical impedance analysis (BIA)
Waist circumference | End of intervention (12 months)
  Waist circumference
Systolic blood pressure | End of intervention (12 months)
  Systolic blood pressure
Diastolic blood pressure | End of intervention (12 months)
  Diastolic blood pressure
Serum leptin | End of intervention (12 months)
  Concentrations of serum leptin
Total cholesterol | End of intervention (12 months)
  Concentrations of serum total cholesterol
Low density lipoprotein (LDL) | End of intervention (12 months)
  Concentrations of serum low density lipoprotein (LDL) cholesterol
Triglycerides | End of intervention (12 months)
  Concentrations of serum triglycerides
Insulin | End of intervention (12 months)
  Concentrations of serum insulin

CONTACTS AND LOCATIONS:
Overall Officials: Jens-Christian Holm, Ph.d., MD, Study Chair — The Children's Obesity Clinic, Department of Pediatrics, Holbæk Hospital, Part of Copenhagen University Hospital
Locations (5):
- Denmark (5):
  - Municipality heath center, Ballerup, Ballerup Municipality, Ballerup
  - Municipality health center, Frederikssund Kommune, Frederikssund, Frederikssund
  - Municipality health center, Guldborgsund, Nykøbing Falster, Guldborgsund
  - Municipality heath center, Lejre, Lejre
  - Municipality heath center, Solrød, Solrød Strand

IPD SHARING:
Plan to Share IPD: Yes
After the results have been published, the aim is to make a depersonalised dataset publicly available on e.g. ClinicalTrials.gov and/or the European Union (EU) Zenodo database (https://zenodo.org/). The final choice will reflect which platform(s) that are compliant with current legislation at that time.
Supporting Information: Study Protocol, SAP
Time Frame: When the results have been published
Access Criteria: Researchers with a protocol for their planned study